CLINICAL TRIAL: NCT03878186
Title: Efficacy Of A Cognitive Behavioral Therapy To Decrease Threat Appraisal In Participants With HIV Infection Initiating Antiretroviral Treatment: Clinical Trial
Brief Title: Efficacy Of A Cognitive Behavioral Therapy To Decrease Threat Appraisal In HIV Participants Initiating Antiretroviral
Acronym: AppraHIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Collaborators: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Responsible Party: Principal Investigator, Jessica Mejía Castrejón, Doctoral student. Staff psychologist, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REF. 2695
Record Dates: First submitted 2019-02-09; First posted 2019-03-18 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: HIV; Threat Appraisal
Keywords: HIV; Threat appraisal; Cognitive behavioral therapy; Antiretroviral-naïve; Challenge appraisal; Affect; Adherence; Quality of life; Anxiety; Depression; Viral load; Loss to follow-up
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (CBT) (Experimental): Cognitive behavioral therapy (CBT). Participants will receive the usual care and 6 sessions of cognitive behavioral therapy
  Interventions: Other: Usual Care (UC); Behavioral: Cognitive Behavioral Therapy (CBT)
- Usual Care (UC) (Other): Participants will receive Usual Care only
  Interventions: Other: Usual Care (UC)

INTERVENTIONS:
Other: Usual Care (UC) — Usual Care: single in-person psycho-educative session with information about HIV, transmission, natural history of the disease, importance of antiretroviral adherence. All the information is based on guidelines and information sheets from InfoVIHt
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive behavioral therapy (CBT): Usual Care + Cognitive-behavioral therapy program intervention (AppraHIV). This intervention involves 7 in-person weekly sessions based on Adjuvant Psychological Therapy centered in three areas: cognitive appraisal, affect and adherence and self-care, everyone with different techniques: cognitive techniques, diaphragmatic breathing, scheduling pleasurable activities, use of pillbox, solving problems, planning for the future, etc. The intervention was manualized (according to Template for Intervention Description and Replication TIDieR), piloted and validated.
  Arms: Cognitive behavioral therapy (CBT)

SUMMARY:
Studies in the field of health and HIV indicate that threat appraisal is associated with poor adherence to treatment, anxiety, poor quality of life, avoidance behavior, less antiretroviral adherence, negative affect, social, instrumental and emotional stress, depression, global distrés, poor subjective health and psychological distres. Most psychological interventions have been oriented to behavioral aspects, leaving aside cognitive aspects such as threat appraisal, so is necessary to investigate psychological treatments and its impact in threat appraisal an in an clinical and psychological outcomes.

Primary objective: To evaluate the efficacy of a cognitive behavioral therapy (CBT) to decrease threat appraisal in comparison with Usual Care (UC) in HIV patients initiating antiretroviral treatment at week 8.

Secondary objectives: To evaluate the effect of a cognitive behavioral therapy intervention compared with Usual Care in HIV patients initiating antiretroviral treatment in the following variables: challenge appraisal, affect (positive and negative), adherence, quality of life, anxiety and depression, HIV viral load and loss to follow-up at weeks 8, 20 and 52.

Exploratory objectives: To assess the threat appraisal cut-off value that predicts favorable outcomes in adherence, virologic suppression, retention in care and adverse events at week 52.

The study is an open label, single center, parallel group clinical trial, in which 50 participants will be randomly assigned using a blocked design to one of the 2 arms: Usual Care (single individual psycho-educative session) or Cognitive Behavioral Therapy (Usual care + 6 sessions of individual Cognitive Behavioral Therapy). The sample will be conformed with 50 adults with HIV, naïve to ARV treatment, starting care at INCMNSZ, who have scores of threat appraisal ≥40 in the CEAT scale, without severe mental disorders or cognitive impairment. We will use independent t test and chi square and intention to treat analysis for the primary outcome, also for secondary outcomes t student for continuous variables, chi square for categorical variables and per protocol analysis in participants adherent to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* HIV diagnosis confirmed
* Naïve to antiretroviral treatment
* Threat appraisal greater than or equal to 40%
* Enrolled at INCMNSZ for medical care
* Be able to read and write
* Willing and able to provide written informed consent

Exclusion Criteria:

* Psychotic symptoms
* Severe depression
* Severe anxiety
* Suicide risk
* Substance dependence
* Cognitive dysfunction
* Psychological or psychiatric treatment within previous 3 months
* Require emergency medical attention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Threat appraisal: Difference in the average scores of threat appraisal at week 8 (continuous) | Measured at baseline and week 8
  Subscale of threat appraisal from HIV/AIDS Stress Scale (EAC-VIH). The subescale of threat appraisal is a validated self-report questionnaire, with 6 items. Participants rate how much they perceived HIV-related problem has damaged different areas (including life goals, self-respect and health) according to likert scale from 1 (no harm) to 5 (extremely harmful). Scores are summed and transformed in percentages. High values indicate worst severity of threat.
Threat appraisal: Proportion of subjects with success (change >54% in threat appraisal at week 8 (nominal binary) | Measured at baseline and week 8
  Subscale of threat appraisal from HIV/AIDS Stress Scale (EAC-VIH). The subescale of threat appraisal is a validated self-report questionnaire, with 6 items. Participants rate how much they perceived HIV-related problem has damaged different areas (including life goals, self-respect and health) according to likert scale from 1 (no harm) to 5 (extremely harmful). Scores are summed and transformed in percentages. High values indicate worst severity of threat.

SECONDARY OUTCOMES:
Challenge appraisal: Difference in the average scores of challenge appraisal | Measured at baseline and weeks 8, 20 and 52
  Subscale of challenge appraisal from HIV/AIDS Stress Scale (EAC-VIH). The subescale of challenge appraisal is a validated self-report questionnaire with 3 items. Participants indicate the extent to which the HIV-problem related provided potential for personal growth, personal challenge or strengthening for a relationship. Challenge appraisal is rated according to 5 Likert scale from 1 (nil potential) to 5 (high potential). Scores are summed and transformed in percentages. High values indicate high potential for growth.
Positive and negative affect: Difference in the average scores of positive and negative affect | Measured at baseline and weeks 8, 20 and 52
  Positive and negative affect Schedule (PANAS): PANAS is a validated self-report measure of affect. This scale has 20 items distributed in 2 scales (positive affect and negative affect) The subjects are instructed to rate the extent to which they experienced each mood state on a 5-point scale (1= very slightly or not at all - 5 = extremely) during the past week. The total score is the sum of the 10 positive items and the 10 negative items. Scores range from 10 to 50 for both set of items. High scores in positive affect indicate high pleasant states. High scores in negative affect indicate high unpleasant states.
Adherence to HIV therapy: Proportion of subjects with adherence >85% | Measured at baseline and weeks 8, 20 and 52
  Questionnaire to evaluate the adherence to HIV therapy (CEAT-VIH). CEAT-VIH is a self-reported questionnaire that assess the level of adherence to antiretroviral therapy. This multidimensional questionnaire has 20 items. Most items are rated using likert scale. The scores range from 17 to 89. Strict adherence = percentile ≥ 85, insufficient adherence = ≤84.
Health related quality of life: Difference in the average scores of quality of life | Measured at baseline and weeks 8, 20 and 52
  Medical Outcomes Study HIV Health Survey (MOS-HIV). MOS-HIV is a self-administered measure of functional status and well-being in HIV patients. It includes 35 items and assesses 10 dimensions. The scores are transformed to a standardized scale ranging from 0% to 100%, where higher scores indicate better quality of life.
Depression and anxiety: Difference in the average scores of depression and anxiety | Measured at baseline and weeks 8, 20 and 52
  Hospital Anxiety and Depression Scale (HAD). HADS is a fourteen ítem scale with 2 scales. Seven of the items evaluate anxiety, and seven evaluate depression. Each scale rage from 0 to 21. Higher scores indicate higher anxiety/depression complains.
Social support: Propotion of subjects with high social support and success in CBT | Measured at baseline and weeks 8, 20 and 52
  Social Support Questionnaire (SSQ-6). The SSQ-6 quantifies the number of social supports, and satisfaction with social support that is available. The satisfaction ratings are on a 6 point scale ranging from 1 (very dissatisfied) to 6 (very satisfied). The score is calculated averaging the satisfaction score ratings. Scores ≥ 5 in satisfaction with social support will be considered as high social support in this investigation.
Viral load: Proportion of subjects with viral supression | Measured at baseline and month 2, 6 and 10
  Changes in RNA viral load. Viral suprression (cv<400copies/ml)
Loss to follow-up. Proportion of subjects with loss to follow-up | Measured at weeks 8, 20 and 52
  Measure of any missing visit (any missing visits = loss to follow-up)
Adverse events: Frequency and severity of adverse events | Intentional evaluation: Every week until week 8 Report of adverse events until week 52
  Intentional detection of adverse events will be done using a checklist designed for this study. Classification of adverse events will be done using a modified version of Color-Risk Psychiatric Triage (CRPT)
Demographic data: Proportion of subjects by subgroups (age, viral load, etc.), with success in CBT. | Measured at week 8, 20 and 52
  Demographic data. Succes: change of 54% in threat appraisal
Change in threat appraisal and challenge appraisal in every group (CBT, UC) | Measured at week 8, 20 and 52
  The subescale of threat appraisal is a validated self-report questionnaire, with 6 items. Participants rate how much they perceived HIV-related problem has damaged different areas (including life goals, self-respect and health) according to likert scale from 1 (no harm) to 5 (extremely harmful). Scores are summed and transformed in percentages. High values indicate worst severity of threat.

OTHER OUTCOMES:
Adherence | Measured at week 52
  Proportion of participants with adherence ≥95% (Pharmacy pick-up)
Viral supression | Measured at month 10
  Proportion of participants with viral suppression (viral load ≤400/ml)
Retention in care | Measured at week 52
  Proportion of participants retained in care (at least 2 clinic visits per year separated by at least 90 days)
Adverse events | Measured at week 52
  Proportion of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Mejía Castrejón, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
No. There is not a plan to make individual participant data IPD available

REFERENCES:
- [Background] Ahrari S, Mohammadpour A, Amouzeshi Z, Agha-Yousefi A. The Relationship between Cognitive Appraisal and Adherence to Medical Regimens in Type 2 Diabetic Patients. J Caring Sci. 2014 Dec 1;3(4):277-85. doi: 10.5681/jcs.2014.030. eCollection 2014 Dec. PMID 25717457
- [Background] Kennedy P, Lude P, Elfstrom ML, Smithson E. Cognitive appraisals, coping and quality of life outcomes: a multi-centre study of spinal cord injury rehabilitation. Spinal Cord. 2010 Oct;48(10):762-9. doi: 10.1038/sc.2010.20. Epub 2010 Mar 9. PMID 20212500
- [Background] Bigatti SM, Steiner JL, Miller KD. Cognitive appraisals, coping and depressive symptoms in breast cancer patients. Stress Health. 2012 Dec;28(5):355-61. doi: 10.1002/smi.2444. Epub 2012 Aug 10. PMID 22888085
- [Background] Nogueda-Orozco MJ, Fresán-Orellana A, Vite-Sierra A, Sánchez-Sosa JJ, Robles-García R. Escala de apreciación cognitiva del VIH/SIDA: Adaptación y evaluación psicométrica en población mexicana. Psicología Iberoamericana, 14; 55-60, 2015.
- [Background] Pakenham K, Rinaldis M. Development of the HIV/AIDS Stress Scale. Psychology and Health, 17(2):203-219, 2002
- [Background] Pakenham KI, Rinaldis M. The role of illness, resources, appraisal, and coping strategies in adjustment to HIV/AIDS: the direct and buffering effects. J Behav Med. 2001 Jun;24(3):259-79. doi: 10.1023/a:1010718823753. PMID 11436546
- [Background] Meade CS, Wang J, Lin X, Wu H, Poppen PJ. Stress and coping in HIV-positive former plasma/blood donors in China: a test of cognitive appraisal theory. AIDS Behav. 2010 Apr;14(2):328-38. doi: 10.1007/s10461-008-9494-x. Epub 2009 Jan 6. PMID 19127424
- [Background] Robles R, Páez F. Estudio sobre la traducción al español y las propiedades psicométricas de las escalas de afecto positivo y negativo (PANAS). Salud mental, 26(1): 69-75, 2003.
- [Background] Remor E. Valoración de la adhesión al tratamiento antirretroviral en pacientes VIH positivo. Psicothema,14 (2): 262-267, 2002.
- [Background] Pena de Leon E, Aguilar Gaytan SS, Suarez Mendoza AA, Reyes Teran G. [A validation of the MOS-HIV quality of life measure in HIV-infected patients in Mexico]. Rev Panam Salud Publica. 2007 May;21(5):313-9. doi: 10.1590/s1020-49892007000400007. Spanish. PMID 17697485
- [Background] Lopez-Alvarenga JC, Vazquez-Velazquez V, Arcila-Martinez D, Sierra-Ovando AE, Gonzalez-Barranco J, Salin-Pascual RJ. [Accuracy and diagnostic utility of the Hospital Anxiety and Depression Scale (HAD) in a sample of obese Mexican patients]. Rev Invest Clin. 2002 Sep-Oct;54(5):403-9. Spanish. PMID 12587414
- [Background] Robles R, Morales M, Jimenez LM, Morales J. Depresión y ansiedad en mujeres con cáncer de mama: el papel de la afectividad y el soporte social. Psicooncología, 6:191-201, 2009.
- [Background] Molina-Lopez A, Cruz-Islas JB, Palma-Cortes M, Guizar-Sanchez DP, Garfias-Rau CY, Ontiveros-Uribe MP, Fresan-Orellana A. Validity and reliability of a novel Color-Risk Psychiatric Triage in a psychiatric emergency department. BMC Psychiatry. 2016 Feb 10;16:30. doi: 10.1186/s12888-016-0727-7. PMID 26860593
- [Derived] Mejia-Castrejon J, Sierra-Madero JG, Belaunzaran-Zamudio PF, Fresan-Orellana A, Molina-Lopez A, Alvarez-Mota AB, Robles-Garcia R. Development and content validity of EVAD: A novel tool for evaluating and classifying the severity of adverse events for psychotherapeutic clinical trials. Psychother Res. 2024 Apr;34(4):475-489. doi: 10.1080/10503307.2023.2239448. Epub 2023 Aug 8. PMID 37552872